CLINICAL TRIAL: NCT06605365
Title: Ophthalmic Solution in Drye Eye Patients
Brief Title: Cross-linked CMC and Silk Proteins in Eye Disease
Status: Completed | Type: Observational
Sponsor: D&V FARMA srl (Industry)
Collaborators: San Giovanni Addolorata Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: COR-TF
Record Dates: First submitted 2024-09-18; First posted 2024-09-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Dry Eye Disease (DED)
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CXC-SP: Subjects affected by dry eye disease are treated with the new ophthalmic solution containing cross-linked CMC (CX-CMC) and Silk Proteins (SP).
  Interventions: Device: CX-HA and CS

INTERVENTIONS:
Device: CX-HA and CS — Sterile Isotonic ophthalmic solution

SUMMARY:
Data analyses and revision of the DED symptoms. A novel ophthalmic solution containing cross-linked CMC (CX-CMC) and Silk Proteins (SP) has been made available on the market.

Both molecules have been widely studied for their viscoelastic and hydrating, and wound healing properties.

This new ophthalmic solution is the first on the market formulated with a CX-CMC and SP.

ELIGIBILITY:
Inclusion Criteria:

* Subjects affected by dry eye disease

Exclusion Criteria:

* know allergies to CX-CMC
* know allergies to SP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data derived from subject affected by dry eye disease and treated with the ophthalmic solution containing CX-CMC and SP will be collected and analysed
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
TBUT | 3 months
  Tear Breakup Time

SECONDARY OUTCOMES:
OSDI | 3 months
  Ocular Surface Disease Index
Wound Healing | 30 hours
  Scratch test performed on cell lines using the "Ibidi Culture-Inserts". The test provides hinds on the ability of a cell line to cover a "wound" created in the monolayer. Results are given as % of the area covered
UV and Blue light absorption | 0 hours
  The ability of the solution to absorb UV and blue light will be evaluated via a spectrophotometer. The outcome will be measured in arbitrary units.

CONTACTS AND LOCATIONS:
Locations (1):
- San Giovanni-Addolorata Hospital, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Padamwar MN, Pawar AP, Daithankar AV, Mahadik KR. Silk sericin as a moisturizer: an in vivo study. J Cosmet Dermatol. 2005 Dec;4(4):250-7. doi: 10.1111/j.1473-2165.2005.00200.x. PMID 17168872
- [Background] Bobadilla AVP, Arevalo J, Sarro E, Byrne HM, Maini PK, Carraro T, Balocco S, Meseguer A, Alarcon T. In vitro cell migration quantification method for scratch assays. J R Soc Interface. 2019 Feb 28;16(151):20180709. doi: 10.1098/rsif.2018.0709. PMID 30958186
- [Background] Tran SH, Wilson CG, Seib FP. A Review of the Emerging Role of Silk for the Treatment of the Eye. Pharm Res. 2018 Nov 5;35(12):248. doi: 10.1007/s11095-018-2534-y. PMID 30397820
- [Background] D'Aloiso MC, Senzolo M, Azzena B. Efficacy and Safety of Cross-Linked Carboxymethylcellulose Filler for Rejuvenation of the Lower Face: A 6-Month Prospective Open-Label Study. Dermatol Surg. 2016 Feb;42(2):209-17. doi: 10.1097/DSS.0000000000000592. PMID 26771686
- [Background] Lee JS, Lee SU, Che CY, Lee JE. Comparison of cytotoxicity and wound healing effect of carboxymethylcellulose and hyaluronic acid on human corneal epithelial cells. Int J Ophthalmol. 2015 Apr 18;8(2):215-21. doi: 10.3980/j.issn.2222-3959.2015.02.01. eCollection 2015. PMID 25938030
- [Background] Song JK, Lee K, Park HY, Hyon JY, Oh SW, Bae WK, Han JS, Jung SY, Um YJ, Lee GH, Yang JH. Efficacy of Carboxymethylcellulose and Hyaluronate in Dry Eye Disease: A Systematic Review and Meta-Analysis. Korean J Fam Med. 2017 Jan;38(1):2-7. doi: 10.4082/kjfm.2017.38.1.2. Epub 2017 Jan 18. PMID 28197326
- [Background] Barabino S, Benitez-Del-Castillo JM, Fuchsluger T, Labetoulle M, Malachkova N, Meloni M, Utheim TP, Rolando M. Dry eye disease treatment: the role of tear substitutes, their future, and an updated classification. Eur Rev Med Pharmacol Sci. 2020 Sep;24(17):8642-8652. doi: 10.26355/eurrev_202009_22801. PMID 32964952
- [Background] Beckman KA. Characterization of dry eye disease in diabetic patients versus nondiabetic patients. Cornea. 2014 Aug;33(8):851-4. doi: 10.1097/ICO.0000000000000163. PMID 24915011